CLINICAL TRIAL: NCT03791606
Title: Risk Factors,PREvention and outComes for Contrast-Induced Acute Kidney Injury in patientS undErgoing Percutaneous Coronary Intervention at Intensive Care Unit：a Single-center Cohort Study(PRECISE-ICU)
Brief Title: Risk Factors,PREvention and OutComes for CI-AKI in PatientS undErgoing PCI at Intensive Care Unit(PRECISE-ICU)
Acronym: PRECISE-ICU
Status: Completed | Type: Observational
Sponsor: Kaiyang Lin (Other)
Responsible Party: Sponsor-Investigator, Kaiyang Lin, Fujian Provincial Hospital, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Other Study IDs: KLin
Record Dates: First submitted 2018-12-31; First posted 2019-01-02 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: CIN

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective, observational study included all consecutively critically ill patients undergoing percutaneous coronary intervention(PCI) at intensive care unit (ICU) in Fujian Provincial Hospital from January 1st 2012 to December 31st 2018. The aim was to determine the incidence,risk factors,prophylactic strategy and outcomes of CI-AKI in critically ill patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients undergoing PCI at ICU

Exclusion Criteria:

* pregnancy
* lactation
* end-stage renal disease (eGFR <15 mL/min/1.73 m2)
* long-term dialysis treatment
* intravascular administration of contrast medium within the last 7 or 3 days postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Critically ill patients undergoing PCI at ICU were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 755 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
CI-AKI | 1 year
  an absolute SCr increase ≥0.3 mg/dL or a relative increase in SCr ≥50% within 48 hours of contrast medium exposure

SECONDARY OUTCOMES:
in-hospital adverse events | 1 year
  congestive heart failure [CHF], bleeding, stroke, reinfarction, stent thrombosis, required renal replacement therapy, length of hospital stay, hospital costs, and mortality

OTHER OUTCOMES:
MACEs for long-term follow up | 1 year
  mortality,stent restenosis, recurrent myocardial infarction, target vessel revascularization,stroke,bleeding,required renal replacement therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial, Fuzhou, Fujian, China